CLINICAL TRIAL: NCT03898869
Title: Measurement of Revascularization Effect Using Near Infrared Spectroscopy in Below the Knee Arteries
Brief Title: Measurement of Revascularization Effect Using NIRS in BTK Arteries
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vilnius University (Other)
Responsible Party: Principal Investigator, Tomas Baltrūnas, Tomas Baltrūnas, Vilnius University
Other Study IDs: BTK-01
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Percutaneous Transluminal Angioplasty; Wound Heal; Ischemic Feet

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Intraoperative NIRS monitoring — Near infrared spectroscopy non invasively used to register changes in tissue oxygen amount during endovascular revascularization

SUMMARY:
Patient with occluded below the knee arteries and chronic limb ischemia Rutherford class V-VI are enrolled.

During endovascular recanalisation procedure changes in tissue oxygen amount is recorded using near infrared spectroscopy (NIRS).

Primary hypothesis - NIRS can be used to determine sufficient amount of blood reaching the ulcered ishemic area.

Secondary hypothesis - NIRS can be useful in detecting early recoil after BTK recanalisation.

ELIGIBILITY:
Inclusion Criteria:

* Critical limb ischemia Rutherford V-VI
* At least one artery below the knee is planned to revascularize

Exclusion Criteria:

* Blood oxygen saturation below 85% because of any comorbidities
* Life expectancy less than 12 months
* Unavoidable amputation above ankle
* Skin diseases preventing the use of NIRS

Ages: 55 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-comers meeting eligibility criteria in VMK hospital, Vascular surgery department.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Increase in oxygen amount sufficient for wound healing | 12 months

SECONDARY OUTCOMES:
Detection of early recoil after BTK revascularization | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Baltrūnas, Principal Investigator — Vilnius University
Locations (1):
- Vilniaus Miesto Klinikinė hospital, Vilnius, Lithuania